CLINICAL TRIAL: NCT05347407
Title: Biochemical Characterization of Parkinson's Disease-related Proteins in the Enteric Nervous System as a Proxy for Pathological Changes in the Brain
Brief Title: Parkinson's Disease Biomarkers in Nerve Cells in the Gut
Acronym: PD-ENS
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-09020813; 1R01NS136423-01A1 (NIH)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: microbiome; Parkinson's; RBD; Alpha Synuclein; enteric nervous system
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients will be provided with a kit and be asked to bring a stool sample to their colonoscopy appointment. Mucosal biopsies will be collected with standard forceps during colonoscopy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control: Healthy Patients
  Interventions: Procedure: Colonoscopy
- Parkinson's Disease: Patients diagnosed with Parkinson's disease
  Interventions: Procedure: Colonoscopy
- At risk for PD: Defined as REM sleep behavior disorder, known genetic risk factor, and/or first degree relatives with PD
  Interventions: Procedure: Colonoscopy
- Dementia with Lewy Bodies: Patients diagnosed with Dementia with Lewy Body Disease
  Interventions: Procedure: Colonoscopy
- Multiple System Atrophy: Patients diagnosed with Multiple System Atrophy
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Patients will be provided with a kit and be asked to bring a stool sample to their colonoscopy appointment. Mucosal biopsies will be collected with standard forceps during colonoscopy. If the physician determines that the patient will need colonoscopy with biopsy as part of their routine clinical care, they will take 6-8 additional biopsies for use in the research study. If the physician determines that the patient will need colonoscopy without biopsy as part of their routine clinical care, they will take 6-8 biopsies for use in the research study only. The collection of additional biopsies will add an estimated two minutes to the whole procedure.

SUMMARY:
Parkinson's disease affects all the nerve cells in the body, including the ones in the gut. The gut contains its own nervous system, the enteric nervous system, and can be thought of as a "second brain". This second brain can reflect what is going on in the actual brain. This study is being done to look for biomarkers, or early indicators of developing Parkinson's disease, in the microbiome and in the gut tissue taken during routine screening colonoscopy. People aged 45 and over who are due for their routine screening colonoscopy are eligible to participate.

DETAILED DESCRIPTION:
Parkinson's disease affects 1 in 100 people over the age of 65, but the time between disease onset and diagnosis can be many months or years. Interestingly, the pathological hallmarks of Parkinson's disease and other synucleinopathies in the brain can also be seen in the nerve cells in the gut. Parkinson's disease may begin in the gut, at least in some people. Unlike the nerve cells in the brain, the nerve cells in the gut are accessible through routine colonoscopy, and so can be obtained by minimally invasive biopsy for the study in the laboratory. In addition, there are links between gut microbes, including bacteria, and the development of Parkinson's disease.

This research study is being done to discover whether the pathology in enteric nerve cells and the types of bacteria in the gut can serve as an indicator of Parkinson's disease. The goal of this research is to develop a biomarker that could help in earlier diagnosis. It also aims to improve the understanding of the link between the gut and brain in Parkinson's disease.

The American Cancer Society recommends screening colonoscopy starting from the age of 45 for the prevention of colon cancer. The study requires only one visit, and study samples will be collected as part of a colonoscopy needed for routine care.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years old
* Parkinson's Disease defined by the modified UK Parkinson's Disease Society Brain Bank criteria, at risk for the development of Parkinson's disease including REM sleep behavior disorder and/or at least one first degree relative with PD or related disorder, and diseases related to Parkinson's disease including the synucleinopathies Lewy Body Dementia and Multiple System Atrophy.
* Baseline Hoehn & Yahr score 1-4
* No contraindications to undergoing screening colonoscopy
* Able to give informed consent for study participation

Exclusion Criteria:

* Clinical features suggestive of a neurodegenerative diagnosis other than synucleinopathy.
* Diagnosis of primary mitochondrial disorder, epilepsy, stroke, multiple sclerosis or other neurodegenerative diseases such as Alzheimer's disease, Progressive Supranuclear Palsy (PSP), and Corticobasal syndrome.
* Significant concomitant medical disease limiting life expectancy to less than 24 months from study inclusion, or significant and serious concomitant medical disease that is poorly controlled
* Signs of active malignant disease or other clinically relevant abnormality on chest x-ray
* Active or untreated gastrointestinal disease
* Inability to temporarily stop anti-platelet agents or other anti-coagulants without significant risk
* Known substance abuse (recent history of abuse of alcohol or other drugs such as barbiturates, cannabinoids and amphetamines) within last 5 years
* Contraindication to colonoscopy or associated anesthesia
* Pregnancy
* In the opinion of the investigator, any other condition regarded as making subject unsuitable for the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with several stages of Parkinson's disease (PD), aged 45 to 75 years old and healthy age-matched control subjects
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical changes in enteric nervous system | A single timepoint will be evaluated on biopsy samples taken from subjects during routine screening colonoscopy.
  The primary objective of the study is to assess the abundance and subcellular distribution of alpha-synuclein and other Parkinson's disease-related proteins in the enteric nervous system of PD patients and healthy controls.

OTHER OUTCOMES:
Exploratory Objective | 12 months
  Exploratory objectives of the study are to examine whether changes in alpha-synuclein and other biomarkers of Parkinson's disease correlate with age and disease progression. We are interested in whether pathology in the gut precedes or mimics the pathology in the brain, and which areas of the gut are most affected by this pathology. We are also interested in whether we can detect pathological changes in alpha-synuclein and other PD biomarkers, including changes in microbiome, at an early disease stage in humans

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Burre, PhD, Principal Investigator — Weill Medical College of Cornell University; Virginia M Gao, MD PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No